CLINICAL TRIAL: NCT02829489
Title: International Audit of Nutrition Care in Patients With FORegut TuMors
Brief Title: International Nutrition Audit in FORegut TuMors
Acronym: INFORM
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Fresenius Kabi (Industry); Nutricia Advanced (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 11111
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Head and Neck Cancer; Esophageal Cancer
Keywords: nutrition; foregut tumors; patient related outcomes; audit
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the current state of nutrition care and patient related outcomes in patients with head, neck and esophageal cancers in North America, Europe and Australia.

DETAILED DESCRIPTION:
The proposed project is a prospective inception cohort study of current nutrition practices of patients with foregut tumors (esophageal and/or head & neck cancer) in cancer care settings in Canada, Europe and Australia. This multi center study will involve a baseline audit of current nutrition practice, followed by repeated audit cycles for up to 6 months from the first time the patient is introduced to the Cancer Care System. Approximately 5-7 Cancer Care settings from Europe, Australia and North America will participate in this audit.

All consecutive consenting patients will be enrolled in the study. As an audit, a formal sample size calculation is not possible, however, we estimate that each of the 5-7 sites will be able to enroll 20 patients over 1 year, with a 6 month follow up, resulting in an estimated sample size of 140-200. All the nutrition care characteristics, patient level descriptors and patient related outcomes will be described using mean and standard deviation or median and inter quantile range based on distributional properties for continuous variables by different locations and cancer care settings. Count with percentages will be used for categorical variables. The effect of route of nutrition, timing of initiation of nutrition intervention, adequacy of nutrition, Patient Generated Subjective Global Assessment (PGSGA) scores and scores of weight, food intake, symptoms and activities & function on survival of the patients will be assessed by univariate and multi-variable Cox regression.

The association of categorical factors such as route of nutrition, timing of initiation of nutrition intervention and so on with the categorical outcomes-complications related to cancer treatment, unplanned readmission and treatment toxicity-will be assessed by chi-square or Fisher exact test, as appropriate. The continuous variables such as PGSGA and other scores will be compared between different categories of the outcomes by t-test or ANOVA as appropriate. Appropriate non-parametric test will be conducted if distributional properties invalidate the use of t-test or ANOVA. The association of continuous variables with continuous outcomes will be assessed by Pearson or Spearman correlation. If necessary, multivariable analyses will be conducted using multiple regression analysis for continuous outcomes and logistic regression for binary outcomes.

Data will be stored in REDCap system housed in a physically and electronically secure data centre at the University of Alberta and is behind the Faculty of Medicine's firewall. REDCap is a secure, web-based application designed exclusively to support data capture for research studies. REDCap provides: 1) an intuitive interface for data entry (with data validation); 2) 128 bit encryption between the data entry client and the server; 3) audit trails for tracking data manipulation and export procedures; 4) automated export procedures for seamless data downloads to common statistical packages (SPSS, Statistical Analysis Software [SAS], Stata, R); 5) procedures for importing data from external sources; and 6) advanced features, such as branching logic, calculated fields and data quality checks.

After this pilot study is completed, we hope to enhance the nutrition evidence in this area by expanding this work to create a prospective registry of nutrition practices and outcomes in patients with foregut tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Head and Neck or Esophageal Cancer and
2. At least 18 yrs age.

Exclusion Criteria:

1. At the time of diagnosis of cancer, if there is no treatment plan due to patient's imminent death OR
2. At the time of diagnosis of cancer, patient's Eastern Cooperative Oncology Score (ECOG) score is ≥ 4

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with head and/or neck cancer or esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Delivery of nutrition intervention | up to a maximum of 6 months
  What is the timing of start of nutrition, adequacy of nutrition and the route of nutrition (oral, enteral and/or parenteral)

SECONDARY OUTCOMES:
Correlation of route of nutrition with outcomes | up to a maximum of 6 months
  Does the route of nutrition (oral, enteral, if enteral either gastric or jejunal or parenteral) correlate with survival, complications related to cancer treatment, unplanned re-admissions, treatment tolerance and treatment toxicity
Correlation of timing of start of nutrition with outcomes | up to a maximum of 6 months
  Does the timing of initiation of nutrition intervention correlate with survival, complications related to cancer treatment, unplanned re-admissions, treatment tolerance and treatment toxicity
Correlation of adequacy of nutrition with outcomes | up to a maximum of 6 months
  Does the adequacy of nutrition intervention correlate with survival, complications related to cancer treatment, unplanned re-admissions, treatment tolerance and treatment toxicity
Correlation of patient generated assessments with outcomes | Baseline, 2, 4 and 6 months
  Does the PGSGA correlate with survival, complications related to cancer treatment, unplanned re-admissions, treatment tolerance and treatment toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Leah Gramlich, MD, FRCP, Principal Investigator — University of Alberta
Locations (7):
- University of California, Davis Medical Center, Sacramento, California, United States
- Australia (2):
  - Chris O Brien Lifehouse & Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
- Canada (2):
  - University of Alberta, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
- Sapienza University, Rome, Italy
- VU University Medical Center, Amsterdam, MB, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Only the aggregate of all anonymous participant data will be shared with the participating sites upon request. The site specific anonymous participant data will be shared with the site upon request. This is detailed in the Data Transfer Agreement with each site.
Supporting Information: CSR
Time Frame: December 2018
Access Criteria: In accordance with the Data Sharing Agreements and contracts with each researcher

REFERENCES:
- [Background] Lees J. Incidence of weight loss in head and neck cancer patients on commencing radiotherapy treatment at a regional oncology centre. Eur J Cancer Care (Engl). 1999 Sep;8(3):133-6. doi: 10.1046/j.1365-2354.1999.00156.x. PMID 10763643
- [Background] Hammerlid E, Wirblad B, Sandin C, Mercke C, Edstrom S, Kaasa S, Sullivan M, Westin T. Malnutrition and food intake in relation to quality of life in head and neck cancer patients. Head Neck. 1998 Sep;20(6):540-8. doi: 10.1002/(sici)1097-0347(199809)20:63.0.co;2-j. PMID 9702542
- [Background] Van Cutsem E, Arends J. The causes and consequences of cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S51-63. doi: 10.1016/j.ejon.2005.09.007. PMID 16437758
- [Background] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Background] Rabinovitch R, Grant B, Berkey BA, Raben D, Ang KK, Fu KK, Cooper JS; Radiation Therapy Oncology Group. Impact of nutrition support on treatment outcome in patients with locally advanced head and neck squamous cell cancer treated with definitive radiotherapy: a secondary analysis of RTOG trial 90-03. Head Neck. 2006 Apr;28(4):287-96. doi: 10.1002/hed.20335. PMID 16287132
- [Background] Arends J, Bodoky G, Bozzetti F, Fearon K, Muscaritoli M, Selga G, van Bokhorst-de van der Schueren MA, von Meyenfeldt M; DGEM (German Society for Nutritional Medicine); Zurcher G, Fietkau R, Aulbert E, Frick B, Holm M, Kneba M, Mestrom HJ, Zander A; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Non-surgical oncology. Clin Nutr. 2006 Apr;25(2):245-59. doi: 10.1016/j.clnu.2006.01.020. Epub 2006 May 12. PMID 16697500
- [Background] Martin L, de van der Schueren MA, Blauwhoff-Buskermolen S, Baracos V, Gramlich L. Identifying the Barriers and Enablers to Nutrition Care in Head and Neck and Esophageal Cancers: An International Qualitative Study. JPEN J Parenter Enteral Nutr. 2016 Mar;40(3):355-66. doi: 10.1177/0148607114552847. Epub 2014 Oct 6. PMID 25288589
- [Background] Rose-Ped AM, Bellm LA, Epstein JB, Trotti A, Gwede C, Fuchs HJ. Complications of radiation therapy for head and neck cancers. The patient's perspective. Cancer Nurs. 2002 Dec;25(6):461-7; quiz 468-9. doi: 10.1097/00002820-200212000-00010. PMID 12464838
- [Background] Howell D, Molloy S, Wilkinson K, Green E, Orchard K, Wang K, Liberty J. Patient-reported outcomes in routine cancer clinical practice: a scoping review of use, impact on health outcomes, and implementation factors. Ann Oncol. 2015 Sep;26(9):1846-1858. doi: 10.1093/annonc/mdv181. Epub 2015 Apr 17. PMID 25888610
- See also: Evidence based practice guidelines for the nutritional management of adult patients with head and neck cancer. Clinical Oncology Society of Australia (COSA). — http://wiki.cancer.org.au/australia/COSA:Head_and_neck_cancer_nutrition_guidelines